CLINICAL TRIAL: NCT01646151
Title: A Study Comparing IOP-Lowering Treatments to Bimatoprost in Patients With Primary Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/OPH/GLA/033
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Results first posted 2014-06-13 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-05

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost; Ganfort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bimatoprost: Bimatoprost-containing eye drops administered in the affected eye(s) at a dose determined by the physician in accordance with standard of care for up to 12 weeks.
  Interventions: Drug: Bimatoprost

INTERVENTIONS:
Drug: Bimatoprost — Bimatoprost-containing eye drops administered in the affected eye(s) at a dose determined by the physician in accordance with standard of care for up to 12 weeks.
  Other Names: LUMIGAN®; GANFORT®

SUMMARY:
An observational study comparing changing from an IOP-lowering treatment to a bimatoprost-containing IOP treatment in primary open-angle glaucoma (POAG) or ocular hypertension (OHT). Visits and treatment are per normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of POAG or OHT
* Previous use of IOP-lowering medication

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with POAG and OHT
Sampling Method: Non-Probability Sample
Enrollment: 2580 (Actual)
Dates: Start 2012-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Dresden, Germany
- Amsterdam, Netherlands

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bimatoprost
Started | 2580
Completed | 2410
Not Completed | 170

BASELINE CHARACTERISTICS:
Arm/Group | Bimatoprost
Number analyzed (Participants) | 2580
Age, Customized [Number; unit: Participants]
  <18 years | 0
  18 to 30 years | 12
  31 to 40 years | 20
  41 to 50 years | 178
  51 to 60 years | 403
  61 to 70 years | 695
  71 to 80 years | 883
  81 to 90 years | 342
  >=91 years | 19
  Missing | 28
Sex/Gender, Customized [Number; unit: Participants]
  Female | 1454
  Male | 1115
  Missing | 11

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP) at Baseline
Description: IOP is a measurement of the fluid pressure inside the eye. IOP was measured in the left and right eyes at Baseline.
Time Frame: Baseline
Population: All patients with data for this outcome measure
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Bimatoprost
Number analyzed (Participants) | 2099
Millimeters of Mercury (mmHg)
  Right Eye | 20.51 (4.32)
  Left Eye (n=2091) | 20.65 (4.54)

2. Secondary Outcome: Physician Evaluation of IOP Lowering in the Study Eye(s)
Description: IOP is a measurement of the fluid pressure inside the eye. Physicians evaluated IOP compared to the target IOP for each patient's study eye(s). The numbers of eyes in each category are presented.
Time Frame: Week 12
Population: All patients with data for this outcome measure
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Bimatoprost
Number analyzed (Participants) | 2375
Number analyzed (Eyes) | 2671
Eyes
  IOP lower than target | 622
  Target IOP reached | 1173
  IOP decreased but target not reached | 467
  IOP increased | 85
  No change | 119
  Data Missing | 205

3. Secondary Outcome: Patient Assessment of Tolerability on a 4-Point Scale
Description: Patient assessment of tolerability was assessed using a 4-point scale (very good, good, moderate, and poor). The numbers of patients in each category are presented.
Time Frame: Week 12
Population: All patients with data for this outcome measure
Measure: Number; unit: Patients
Arm/Group | Bimatoprost
Number analyzed (Participants) | 2347
Patients
  Very Good | 1127
  Good | 1070
  Moderate | 80
  Poor | 70

4. Secondary Outcome: Physician Assessment of Tolerability on a 4-Point Scale
Description: Physician assessment of tolerability was assessed using a 4-point scale (very good, good, moderate, and poor). The numbers of patients in each category are presented.
Time Frame: Week 12
Population: All patients with data for this outcome measure
Measure: Number; unit: Patients
Arm/Group | Bimatoprost
Number analyzed (Participants) | 2369
Patients
  Very Good | 1212
  Good | 1059
  Moderate | 74
  Poor | 24

5. Secondary Outcome: Physician Assessment of Patient Compliance Compared to Previous Therapy
Description: Physician assessment of patient compliance compared to previous therapy was assessed on a 3-point scale (better, equal, and worse). The numbers of patients in each category are presented.
Time Frame: Week 12
Population: All patients with data for this outcome measure
Measure: Number; unit: Patients
Arm/Group | Bimatoprost
Number analyzed (Participants) | 2113
Patients
  Better | 875
  Equal | 1151
  Worse | 51
  Not Applicable | 36

6. Secondary Outcome: Percentage of Patients Who Discontinue Treatment With Bimatoprost-Containing Eye Drops Prior to 12 Weeks of Treatment
Description: Patients who discontinue treatment with bimatoprost-containing eye drops prior to 12 weeks of treatment was assessed as Yes or No.
Time Frame: 12 Weeks
Population: All patients
Measure: Number; unit: Percentage of Patients
Arm/Group | Bimatoprost
Number analyzed (Participants) | 2580
Percentage of Patients | 6.6

7. Secondary Outcome: Percentage of Patients Who Continue Treatment With Bimatoprost-Containing Eye Drops
Description: Patients who will continue treatment with bimatoprost-containing eye drops after 12 weeks of treatment was assessed as Yes or No.
Time Frame: Week 12
Population: All patients
Measure: Number; unit: Percentage of Patients
Arm/Group | Bimatoprost
Number analyzed (Participants) | 2580
Percentage of Patients | 85.8

8. Primary Outcome: IOP at Week 12
Description: IOP is a measurement of the fluid pressure inside the eye. IOP was measured in the left and right eyes at Week 12.
Time Frame: Week 12
Population: All patients with data for this outcome measure
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Bimatoprost
Number analyzed (Participants) | 2099
Millimeters of Mercury (mmHg)
  Right Eye | 15.78 (2.85)
  Left Eye (n=2091) | 15.87 (3.19)

ADVERSE EVENTS:
Description: All enrolled patients were used to assess adverse events (AEs) and serious adverse events (SAEs).
Arm/Group | Bimatoprost
Serious Adverse Events (participants affected / at risk) | 0/2580
Other Adverse Events (participants affected / at risk) | 450/2580
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost (N=2580)
Conjunctival Hyperaemia (Eye disorders) | 292
Eye Irritation (Eye disorders) | 158

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.